CLINICAL TRIAL: NCT03591965
Title: An Open-label Phase 2 Trial of Dual TORC1/TORC2 Inhibitor ATG-008 in HBV+ Advanced Hepatocellular Carcinoma (HCC) Subjects Who Have Received at Least One Prior Line of Systemic Therapy (TORCH)
Brief Title: Dual TORC1/TORC2 Inhibitor ATG-008 (CC-223) in HBV Positive Advanced Hepatocellular Carcinoma (HCC) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the adjustment of clinical research and development strategy，sponsor decided to terminate the study
Sponsor: Antengene Therapeutics Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-008-HCC-001
Record Dates: First submitted 2018-06-20; First posted 2018-07-19 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-008 (Experimental): To enroll approximately 40 hepatitis B virus (HBV) positive, unresectable HCC subjects who have previously received at least one prior line of systemic therapy. Among which, approximately 20 subjects will receive oral ATG-008 at an initial dose of 45 mg, once daily (QD) and another approximately 20 subjects will receive oral ATG-008 at an initial dose of 20 mg, twice daily (BID). The pharmacokinetic (PK) samples will be collected from 10 subjects each in the two dose groups.
  Interventions: Drug: ATG-008

INTERVENTIONS:
Drug: ATG-008 — Approximately 20 subjects will receive oral ATG-008 at an initial dose of 45 mg/QD and another 20 subjects will receive oral ATG-008 at an initial dose of 20mg/BID for 28 days each cycle.

SUMMARY:
This is an Asian multi-regional clinical trial (MRCT) in which ATG-008 will be administered orally to hepatitis B positive (HBV+) HCC subjects who have received at least one prior line of systemic therapy. It is designed as an open-label phase 2 trial evaluating the pharmacokinetics (PK), safety, tolerability and efficacy of oral ATG-008 administered daily until the radiologic disease progression (according to RECIST 1.1) or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged from 18 to 70 years (inclusive) at the time when the ICF is signed.
2. Confirmed diagnosis of HCC.
3. Unresectable stage B or C HCC according to the Barcelona Clinic Liver Cancer (BCLC) staging.
4. HBV positive by serum test.
5. Received at least one prior line of systemic therapy.
6. ECOG performance status score of 0 or 1.
7. Satisfactory serum chemistry results
8. Adequate bone marrow function
9. Child-Pugh A without encephalopathy.
10. All subjects who participated in the study had to take reliable contraceptive measures within the trial and 3 months of after the trial.

Exclusion Criteria:

1. Symptomatic central nervous system metastases.
2. Locoregional HCC therapy, systemic chemotherapy, hormonal therapy or investigational therapy within 4 weeks prior to Screening.
3. Life expectancy of less than 3 months.
4. Prior therapy with mTOR inhibitors.
5. Prior organ transplant.
6. Persistent diarrhea or malabsorption.
7. Clinically significant bleeding.
8. Known history of human immunodeficiency virus (HIV) infection.
9. Uncontrolled intercurrent illness.
10. Any condition that confounds the ability to interpret data from the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 - Day 15
  Peak Plasma Concentration (Cmax)
AUC | Day 1 - Day 15
  Area under the plasma concentration versus time curve (AUC)
The incidence of treatment emergent adverse events (TEAEs) & SAE assessed by CTCAE v4.03 | 365 DAYS
  The treatment emergent adverse events (TEAEs) & SAE case No. in total subject No.
ORR | 365 DAYS
  Percentage of subjects with PR, or CR

SECONDARY OUTCOMES:
OS | 365 DAYS
  Kaplan-Meier estimate of Overall Survival
TTP | 365 DAYS
  The time from the first dose date until disease progression
PFS | 365 DAYS
  The time from the first dose date until disease progression or death from any cause
DCR | 365 DAYS
  The percentage of subjects with CR, or PR or stable disease (SD)
DOR | 365 DAYS
  The time from the criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented
TTR | 365 DAYS
  The time from the first dose date to the first documentation of response of PR or better.
6, 9 and 12 month of survival rate | 365 DAYS
  Percentage of patients alive

OTHER OUTCOMES:
Potential biomarkers in plasma and tumor tissues | 365 DAYS
  The changes in potential biomarkers including but not limited to TORC1/TORC2 activity in peripheral blood samples and tumor tissue following treatment with ATG-008
Additional metabolites of ATG-008 in plasma and urine | Day 1 - Day 15
  Additional metabolites of ATG-008 in plasma and urine, and the extent of their urinary excretion/clearance

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Xie, PhD, Study Director — Medical Monitor
Locations (30):
- China (19):
  - Oncology Hospital of Haerbin Medical University, Harbin, Heilongjiang
  - China People PLA 81 Hospital, Nanjing, Jiangsu
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The first Hospital of Jilin University, Changchun
  - Hunan Province Oncology Hospital, Changsha
  - Daping Hospital, Chongqing
  - The first hospital of Chongqing medical university, Chongqing
  - Xiehe Hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital of Nanfang Medical University, Guangzhou
  - The first affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Province Oncology Hospital, Hangzhou
  - The first affiliated hospital of Anhui medical university, Hefei
  - The second affiliated hospital of Anhui medical university, Hefei
  - The first affiliated hospital of Guangxi Medical University, Nanning
  - Oncology Hospital of Fudan University, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - General Hospital of the Northern War Zone of the Chinese People's Liberation Army, Shenyang
  - Tangdu Hospital of China PLA fourth medical university, Xi'an
- South Korea (6):
  - Dong-A University Hospital, Busan
  - Pusan National Univ. Hospital, Busan
  - Kyungpook National Univ. Hospital, Daegu
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkuo, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03591965/Prot_SAP_000.pdf